CLINICAL TRIAL: NCT06663397
Title: The Effects Of Laughter Yoga-Supported Childbirth Preparation Training On Traumatic Birth Perception, Fear Of Birth, Prenatal Depression, And Attachment: A Randomized Controlled Study
Brief Title: Laughter Yoga's Impact on Traumatic Childbirth Preparation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, İlknur Münevver Gönenç, Assoc. Prof. Dr., Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ankara U
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Maternal Distress; Prenatal Stress; Pregnancy Related
Keywords: Perception of Traumatic Birth; Fear of Childbirth; Prenatal Depression; Prenatal Attachment; Laughter Yoga; Childbirth Preparation Training
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: A single-center parallel-group randomized controlled trial study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Laughter Yoga-Supported Childbirth Preparation Training) (Experimental): Similar to the control group, the training will be conducted by the researcher, covering the same content as the standard childbirth preparation training. However, in addition to this, the experimental group will participate in Laughter Yoga sessions lasting 45 minutes each week for a total of 4 sessions. These sessions will include 30 minutes of laughter and breathing exercises, followed by 15 minutes of laughter meditation and relaxation
  Interventions: Other: Laughter Yoga; Other: Standard Childbirth Preparation Training
- Control Group (Standard Childbirth Preparation Training) (Active Comparator): The sessions will be conducted in groups of 8 participants. Various educational materials, including visual aids, will be used, and the training will involve presentations, direct instruction, video displays, and question-and-answer sessions.
  Interventions: Other: Standard Childbirth Preparation Training

INTERVENTIONS:
Other: Laughter Yoga — Laughter Yoga sessions lasting 45 minutes each week for a total of 4 sessions. These sessions will include 30 minutes of laughter and breathing exercises, followed by 15 minutes of laughter meditation and relaxation
  Arms: Experimental Group (Laughter Yoga-Supported Childbirth Preparation Training)
Other: Standard Childbirth Preparation Training — the sessions will be conducted in groups of 8 participants. Various educational materials, including visual aids, will be used, and the training will involve presentations, direct instruction, video displays, and question-and-answer sessions

SUMMARY:
This study will be conducted as a single-center, parallel-group, randomized controlled intervention trial to determine the effects of birth preparation training supported by laughter yoga on the perception of traumatic birth, fear of birth, prenatal depression, and attachment in primiparous women. The research population will consist of pregnant women who attend the Pregnancy Clinic of the Department of Obstetrics and Gynecology at Cebeci Medical Faculty, Ankara University. The study will involve two groups: the first group will receive birth preparation training supported by laughter yoga, while the second group will receive standard birth preparation training. A total of 68 pregnant women, 34 in each group, are planned to participate in the study. Data will be collected using the Introductory Information Form, Traumatic Birth Perception Scale, Prenatal Self-Assessment Scale Fear of Birth Subscale, Edinburgh Depression Scale, and Prenatal Attachment Inventory. These instruments will be administered to the participants three times: before the training, immediately after the training, and one month later. The research data will be analyzed using the Statistical Package for Social Sciences (SPSS) version 24. Descriptive statistics (number, percentage, mean, standard deviation, minimum, and maximum values) will be used for data analysis. Independent samples t-test will be employed for comparisons between two independent groups, paired samples t-test will be used for repeated measures, one-way ANOVA will be used for comparisons among more than two groups, and Pearson correlation analysis will be applied for the relationship between two quantitative variables.

When data do not follow a normal distribution, the Mann-Whitney U test will be used for comparisons between two independent groups, the Wilcoxon signed-rank test will be used for repeated measures, the Kruskal-Wallis test will be used for comparisons among more than two groups, and Spearman correlation analysis will be used for the relationship between two quantitative variables. The reliability of the scales used in the study will be determined using Cronbach's alpha coefficient. Statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older.
* Pregnant individuals between 20-26 weeks of gestation (Childbirth preparation training should begin by the 20th week of pregnancy according to the recommendations of the Turkish Ministry of Health, and since the training is planned to last 4 weeks, participants will be recruited before entering the third trimester).
* First-time pregnancies.
* Individuals who understand, speak, and can read and write in Turkish.
* Women who consent to participate in the study.

Exclusion Criteria:

* Women with high-risk pregnancies (such as placenta previa, history of antepartum bleeding, ruptured membranes, preeclampsia, hypertension, diabetes, or other medical conditions, intrauterine growth restriction, multiple pregnancies, fetal anomalies, or any contraindications for normal vaginal delivery, substance or alcohol dependence, chronic illnesses, etc.).
* Individuals diagnosed with psychiatric disorders.
* Those who have received psychotherapy or medication within the last six months prior to the study.
* Pregnant women with prior training or experience in cognitive awareness-based or mind-body methods.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant Women
Enrollment: 68 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Traumatic Birth Perception | It will be administered three times: before the training, immediately after, and one month later.
  • Traumatic Birth Perception Scale: Developed by Yalnız et al. (2016) to assess the level of traumatic birth perception among women of reproductive age, this scale consists of 13 items related to feelings of anxiety, fear, and worry when thinking about childbirth. Scoring ranges from 0 to 10 for each item, with a total possible score of 0 to 130. Higher scores indicate a greater perception of traumatic birth. The Cronbach's alpha reliability coefficient for this scale is 0.89 (Yalnız et al., 2017).
Birth Fear | It will be administered three times: before the training, immediately after, and one month later.
  • Prenatal Self-Assessment Scale Birth Fear Subscale: This scale, developed by Lederman (1979), evaluates pregnant women's adjustment to motherhood. The Turkish reliability and validity study was conducted by Beydağ and Mete (2008). The Birth Fear Subscale consists of 10 items, with possible scores ranging from 10 to 40. Higher scores indicate greater fear of childbirth. The Cronbach's alpha reliability coefficient for this subscale is reported as 0.79 in Lederman's study and 0.84 in Beydağ and Mete's study.
Prenatal Attachment | It will be administered three times: before the training, immediately after, and one month later.
  • Prenatal Attachment Inventory (PBE): Developed by Müller (1993) and adapted to Turkish by Yılmaz and Beji (2013), this 21-item scale assesses emotional experiences and attachment levels during pregnancy. Scores range from 21 to 84, with higher scores indicating stronger attachment. The Cronbach's alpha for this scale is 0.84 (Yılmaz & Beji, 2013), and it will be administered at the same intervals.
Prenatal Depression | It will be administered three times: before the training, immediately after, and one month later.
  • Edinburgh Depression Scale: Developed by Cox et al. (1987), this scale assesses the risk, level, and severity of postpartum depression. The Turkish validity and reliability study was conducted by Engindeniz et al. (1996), with an internal consistency coefficient of 0.79. The scale consists of 10 items rated on a 4-point Likert scale. Although designed for postpartum assessment, it will be used during pregnancy. The Cronbach's alpha coefficients for the three trimesters were 0.82, 0.83, and 0.84, respectively (Bergin et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Gönenç, Assoc. Prof. Dr., Study Chair — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be shared when requested and necessary.